CLINICAL TRIAL: NCT01001481
Title: Clinical Audit and Feedback Program to Determine Risk for Medication Adherence in Outpatients Diagnosed With Schizophrenia in Australia
Brief Title: Schizophrenia Treatment Adherence Investigation (STAI)
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR013822
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Treatment review; Schizophrenia; Observational; Prospective studies; Australia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Risk status for medication adherence

INTERVENTIONS:
Other: Risk status for medication adherence — Examination of risk status for medication adherence in a cohort of Australian patients diagnosed with schizophrenia

SUMMARY:
The primary objective of this treatment review and feedback program is to quantify the risk status for medication adherence in a cohort of Australian patients diagnosed with schizophrenia.

DETAILED DESCRIPTION:
The primary objective of this treatment review and feedback program is to quantify the risk status for medication adherence in a cohort of Australian patients diagnosed with schizophrenia. Observational study - no study drug administered

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV
* Currently treated in an outpatient clinic
* Able to provide informed consent
* Concurrent enrolment in clinical trials is acceptable
* Have completed all questions on the Drug Attitude Inventory (DAI-10) and Medication Adherence Rating Scale (MARS) survey

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure is the Clinical Assessment of Adherence as rated by the Investigators | 6 months, 12 months

SECONDARY OUTCOMES:
Clinical exacerbations (worsening of symptoms) | 6 mths, 12 mths
Medication changes | 6 mths, 12 mths

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd